CLINICAL TRIAL: NCT03888287
Title: Parkinson's Disease Inpatient Clinical Knowledge and Management
Acronym: PICK
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was put on hold due to COVID and never reopened
Sponsor: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00006159
Record Dates: First submitted 2018-08-01; First posted 2019-03-25 (Actual); Results first posted 2023-03-16 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-03

CONDITIONS: Parkinson Disease
Keywords: PICK study; Impact of Watch Rx
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: The WatchRx is a smartwatch worn on the patient's wrist which receives alerts and notifications for medication administration scheduling as well as intervention messages from a App to the caregiver
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Retrospective Phase (Experimental): Patients with Parkinson disease before completion of the Parkinson's Disease Inpatient Clinical Knowledge and Management Program.
  Interventions: Device: Watch Rx system
- Prospective Phase-Watch Rx system (Experimental): Patients after completion of the Parkinson's Disease Inpatient Clinical Knowledge and Management Program who are also assigned to a WatchRx system
  Interventions: Device: Watch Rx system; Other: Parkinson's Disease Inpatient Clinical Knowledge and Management Program
- Retrospective Phase - Clinicians (Experimental): Clinicians, including physician's assistant, advanced practice nurses, staff nurses, nurse educators, case managers, dietitians pharmacists physical therapist and occupational therapist before completion of the Parkinson's Disease Inpatient Clinical Knowledge and Management Program.
  Interventions: Other: Parkinson's Disease Inpatient Clinical Knowledge and Management Program
- Prospective Phase - Clinicians (Experimental): Clinicians, including physician's assistant, advanced practice nurses, staff nurses, nurse educators, case managers, dietitians pharmacists physical therapist and occupational therapist after completion of the Parkinson's Disease Inpatient Clinical Knowledge and Management Program.
  Interventions: Other: Parkinson's Disease Inpatient Clinical Knowledge and Management Program

INTERVENTIONS:
Device: Watch Rx system — The Watch Rx system consists of a Watch Rx smartwatch, Watch Rx application and a WatchRx Web Interface. The Watch Rx smartwatch will be worn on the patient's wrist. The smart watch will send alerts to the caregivers through the Watch Rx app when it is time to administer the medication. The Web Interface will be used to store the medical documentations
  Arms: Prospective Phase-Watch Rx system; Retrospective Phase
Other: Parkinson's Disease Inpatient Clinical Knowledge and Management Program — Parkinson's Disease Inpatient Clinical Knowledge and Management Program educates clinical staff and measures difference in knowledge of medication adherence and compliance for hospitalized Parkinson's Disease patients
  Arms: Prospective Phase - Clinicians; Prospective Phase-Watch Rx system; Retrospective Phase - Clinicians

SUMMARY:
This study will focus on patients with Parkinson's Disease in the adult inpatient units of Hackensack University Medical Center. We are measuring the effect of a Parkinson's Disease Inpatient Clinical Knowledge and Management Program on adherence to Parkinson's Disease medication using a Parkinson's Disease Identification Wrist Band, smartwatch and medication schedule card

DETAILED DESCRIPTION:
Parkinson's Disease (PD), the second-most common neurodegenerative disorder and is ranked the fourteenth leading cause of death. PD prevalence rate in the United States is estimated to be approximately 0.3% and is ranked the fourteenth leading cause of death (CDC, 2013). Depending on the methodology, the national prevalence data on PD is varied and insufficient. PD is projected to increase by 4% to 5% in age 65 and over 85 years respectively and is associated with a high economic burden exceeding $14.4 billion per year.

Admission to the hospital is identified as a major risk factor due to imprecise timing of medication administration, disruption of sleep pattern, dietary changes, and unfamiliarity of the hospital environment which all contribute to the exacerbation of PD symptoms. Parkinson's disease Foundation, 2015). Hospital length of stay for patients with PD is 1.45 times higher in comparison to non- PD patients.

A study by Chou et al., (2011) involving 51 worldwide National Parkinson Foundation Centers found 94% of centers were not confident in the care and knowledge hospital professionals provided specific to: PD medications, complex drug interactions, contraindications and precise timing of medication administration. Hospital co-morbidities could be improved or prevented by adjustment of PD medication and medication adherence, critical in decreasing hospital length of stay.

The retrospective phase will be a data collection of adult patients admitted with a primary and secondary diagnosis of Parkinson's disease during January - June 2015 (6 month period). There will be 150 patients selected by the principal investigator(s) from chart review. In addition, the clinicians chosen for the study will complete a Parkinson's Disease Knowledge Assessment Survey.

The prospective phase will begin after completion of the Parkinson's Disease Inpatient Clinical Knowledge and Management Program for staff nurses, advanced practice nurses (APN), nursing assistants, patient care technicians, case managers, adult inpatient physician assistants, pharmacists, occupational therapists, physical therapists, nurse educators, and dietitians. There will be 150 patients selected from the adult inpatient units by the principal investigator(s) that meet the inclusion criteria and confirm through an informed consent that they will participate in the study.

The selected patients will be registered in a WatchRx interface via website URL by the Principal Investigator(s) and the Transition of Care(TC) Pharmacist and required to wear a Watch Rx smartwatch for the duration of their hospitalization. The Watch Rx Interface will store all medical information, necessary treatments, and daily clinical care for the patient which is synchronized to the smartwatch on the patient's wrist. The smartwatch will send alerts to the patient's assigned nurse's iPad through a Watch Rx app for medication administration, missed PD medications, battery conditions, and enables messaging between the primary nurse and the patient.

The WatchRx smartwatch will remind when it is time to take the medication. If the Parkinson's Disease medication is not administered, it sends missed medication reminder alerts to the nurse. For fixed time medication, the reminder is every 3 minutes up to 10 minutes.

During the prospective phase, the research team will collect data from multiple sources such as the Watch Rx system, EPIC Hyperspace, and Case Report forms over a 6 month study period. The data will be calculated by using statistical analysis for the continuous variables and categorical variables identified from the collection of data. All study data will be imported into SAS software where data programming will be utilized to flag and generate queries on out-of-range data issues until they are resolved. All analysis will be performed using SAS version 9.4 (SAS Institute Inc. Cary, North Carolina, USA Data will be handled in a confidential manner to meet mandated IT Security standards and to prevent loss of privacy. All electronic files will be stored in an encrypted and password-protected database on a secure medical center server. Only co-investigators, advanced practice nurses, and the data coordinator who contact the subjects will have access to information linked to subject identifiers.

This study will improve timely administration of medications to PD patients. Patients enrolled in the study will have direct monitoring of their medication compliance and adherence. Patients participating in the registry will be gain information from the current research and possibly create a support group amongst themselves. This study will improve knowledge of Parkinson's disease amongst clinicians and better medication management of PD patients

ELIGIBILITY:
Inclusion Criteria:

* Adult patients diagnosed with primary and secondary diagnosis of Parkinson's disease
* Patient 22 years old and older
* Patients admitted to inpatient units
* Patient who are verbally informed and agree to participate in the study

Exclusion Criteria:

* Patients less than or equal to 21 years of age
* Patients who refuse to wear the PD wrist band.
* Patients who verbally refuse enrollment in the PD registry.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 477 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2022-01-03 (Actual); Study Completion 2022-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Azmi Hooman, MD, Principal Investigator — Hackensack Meridian Health; Mohammed Quadri, MD, MBA, Principal Investigator — Hackensack Meridian Health
Locations (1):
- Hackensack University Medical Center, Hackensack, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Retrospective Phase: Patients with Parkinson's disease before completion of the Parkinson's Disease Inpatient Clinical Knowledge and Management Program.
- Retrospective Phase - Clinicians: Clinicians, including physician's assistants, advanced practice nurses, staff nurses, nurse educators, case managers, dietitians pharmacists physical therapists, and occupational therapists before completion of the Parkinson's Disease Inpatient Clinical Knowledge and Management Program.
- Prospective Phase - Clinicians: Clinicians, including physician's assistants, advanced practice nurses, staff nurses, nurse educators, case managers, dietitians pharmacists physical therapists and occupational therapists after completion of the Parkinson's Disease Inpatient Clinical Knowledge and Management Program.
Period: Overall Study
Arm/Group | Retrospective Phase | Prospective Phase-Watch Rx System | Retrospective Phase - Clinicians | Prospective Phase - Clinicians
Started | 131 | 0 | 266 | 80
Completed | 131 | 0 | 266 | 80
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No one was enrolled in the patient prospective phase.
Groups:
- Total: Total of all reporting groups
Arm/Group | Retrospective Phase | Prospective Phase-Watch Rx System | Total
Number analyzed (Participants) | 131 | 0 | 131
Age, Customized [Mean (Standard Deviation); unit: years] — Prospective enrollment was unable to occur due to the COVID-19 pandemic and restrictions.
  years | 76 (14.4) |  | 76 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Information/demographics of clinicians was never collected.
  Participants
    Female | 54 | 0 | 54
    Male | 77 | 0 | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Demographic data was never collected on clinicians.
  Participants
    Hispanic or Latino | 23 | 0 | 23
    Not Hispanic or Latino | 107 | 0 | 107
    Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Demographic data was never collected on clinicians.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 4 | 0 | 4
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 4 | 0 | 4
    White | 106 | 0 | 106
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 17 | 0 | 17
Region of Enrollment [Number; unit: participants]
  United States | 131 |  | 477

OUTCOME MEASURES:

1. Primary Outcome: Clinician's Parkinson's Disease Knowledge Assessment Survey Scores
Description: Clinician's Parkinson's Disease Knowledge Assessment Survey scores before and after the Parkinson's Disease Inpatient Clinical Knowledge and Management Program.
  A 20-question survey was administered to PD clinicians for a group measurement of PD knowledge. Scores ranged from 0 - 100% and reflected the percentage of clinicians who correctly answered the question. If 70% or more clinicians correctly answered the question, the group was considered knowledgeable on that topic; if <70% of clinicians responded incorrectly, they were considered not knowledgeable on the information that the question assessed. Survey questions addressed three PD areas: 1) medication/treatment, 2) symptoms/diagnosis, and 3) epidemiology/pathophysiology.
Time Frame: 6 months
Population: Number of clinicians that completed the pre and post intervention surveys
Measure: Mean (Full Range); unit: average knowledge score
Groups:
- Clinicians' Knowledge Before Educational Intervention: Average clinician's participant PD score before educational intervention
- Clinicians' Knowledge After Educational Intervention: Average clinician's participant PD score after educational intervention
Arm/Group | Clinicians' Knowledge Before Educational Intervention | Clinicians' Knowledge After Educational Intervention
Number analyzed (Participants) | 266 | 80
average knowledge score | 68.50 [0 to 100] | 78.75 [0 to 100]

2. Secondary Outcome: Number of PD Medications Administered on Time (15 Minute Window)
Description: The number of Parkinson's Disease (PD) medications administered within the 15-minute timeframe at baseline
Time Frame: within 15 minutes post PD medication administration time
Population: No patients were enrolled in the study after clinician education
Measure: Number; unit: number of PD meds administered in 15 min
Units Other Than Participants: Number of scheduled PD medications
Groups:
- Retrospective Patient Outcomes: The number of Parkinson's Disease (PD) medical administration administered within 15 minutes of the scheduled time.
Arm/Group | Retrospective Patient Outcomes
Number analyzed (Participants) | 131
Number analyzed (Number of scheduled PD medications) | 2454
number of PD meds administered in 15 min | 678

3. Secondary Outcome: Number of Patients With Contraindicated Medications Administered.
Description: Measure the number of patients who were adminstered contraindicated medications
Time Frame: 6 months
Population: No patients were enrolled in the study after clinician education
Measure: Count of Participants; unit: Participants
Groups:
- Retrospective Patient Outcomes: Parkinson's Disease (PD) patient outcomes before clinicians received PD education
Arm/Group | Retrospective Patient Outcomes
Number analyzed (Participants) | 131
Participants | 21

4. Secondary Outcome: Number Patients With Falls, Falls With Injury, Positive CAM/Mini-cog
Description: The number of falls, number of falls with injury, and number of patients with positive Confusion Assessment Method (CAM)/Mini-Cog scores) in hospitalized patients.
  Mini-cog is performed on all admitted patients 65 years and older and is a quick screening for "cognitive vital sign" and early dementia detection. The scale classifies patients as being positive or negative for dementia.
  The Confusion Assessment Method (CAM) is performed on all adult admissions at the time of admission with reporting 1) every shift if the first test is positive, or 2) daily if the first test is negative. It improves the detection and recognition of delirium accurately and quickly in clinical and research settings. CAM is documentation of observed patient behavior during brief, structured interviews according to classification of positive or negative for dementia. There are no numerical (minimum or maximum) values assigned.
Time Frame: 6 Months
Population: Patients were not enrolled after clinical education
Measure: Count of Participants; unit: Participants
Arm/Group | Retrospective Patient Outcomes
Number analyzed (Participants) | 93
Participants
  Number of falls | 1
  Number of falls with injury | 0
  Number of patients with positive CAM scores | 47
  Number of patients with abnormal mini-cog scores | 45

5. Secondary Outcome: Length of Stay in Hospitalized Parkinson's Disease Patients.
Description: Average length of stay in hospitalized Parkinson's Disease patients
Time Frame: 6 months
Population: Patients were not enrolled after clinical education
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Retrospective Patient Outcomes
Number analyzed (Participants) | 131
days | 6.1 (6.6)

6. Secondary Outcome: Number of PD Medications Administered on Time (Within 15 Minute Window)
Description: Track the difference that the WatchRx system has on scheduled PD medication administration time versus actual PD medication administration time
Time Frame: 15 minutes post assigned medication administration time.
Population: No patients were enrolled for the WatchRX system
Groups:
- Prospective Patient Outcomes (WatchRx): Parkinson's Disease (PD) patient outcomes during implementation of the WatchRX system
Arm/Group | Prospective Patient Outcomes (WatchRx)
Number analyzed (Participants) | 0

7. Secondary Outcome: Number of PD Medication Errors After Using the WatchRX System
Description: The number of contraindicated medications administered to Parkinson's disease patients after using the WatchRX system
Time Frame: 6 Months
Population: No patients were enrolled in the WatchRX system
Arm/Group | Prospective Patient Outcomes (WatchRx)
Number analyzed (Participants) | 0

8. Secondary Outcome: Number of Falls, Falls Within Injury, Positive CAM Scores, and Positive Mini-Cog Scores After Using the WatchRX System
Description: The number of falls, number of falls with injury, number of positive CAM scores, and number of positive Mini-Cog scores after using the WatchRX system.
Time Frame: 6 months
Population: No patient enrollment into the WatchRX system
Arm/Group | Prospective Patient Outcomes (WatchRx)
Number analyzed (Participants) | 0

9. Secondary Outcome: Length of Stay With the WatchRx System
Description: Parkinson's disease patients' length of stay after using the WatchRx system
Time Frame: 6 months
Population: No patients were enrolled into the WatchRX system
Arm/Group | Prospective Patient Outcomes (WatchRx)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 6 months for patient and clinician participants in the Retrospective Phase. Duration of the educational intervention including pre and post-surveys for clinicians in the Prospective Phase, overall duration 5 months
Description: This study was a non-interventional survey-based study. No all-cause mortality was anticipated and none occurred. No Serious adverse events were anticipated and none occurred. No other adverse events were anticipated or occurred.
Groups:
- Retrospective Phase - Watch Rx System: Patients with Parkinson disease before completion of the Parkinson's Disease Inpatient Clinical Knowledge and Management Program.
- Prospective Phase - Watch Rx System: Patients after completion of the Parkinson's Disease Inpatient Clinical Knowledge and Management Program who are also assigned to a WatchRx system
Arm/Group | Retrospective Phase - Watch Rx System | Prospective Phase - Watch Rx System | Retrospective Phase - Clinicians | Prospective Phase - Clinicians
All-Cause Mortality (participants affected / at risk) | 0/131 | 0/0 | 0/266 | 0/80
Serious Adverse Events (participants affected / at risk) | 0/131 | 0/0 | 0/266 | 0/80
Other Adverse Events (participants affected / at risk) | 0/131 | 0/0 | 0/266 | 0/80

LIMITATIONS AND CAVEATS:
Prospective enrollment did not occur due to the COVID-19 pandemic, patients were not admitted for elective surgeries. Results of the clinician education were only reported in aggregate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-09): https://cdn.clinicaltrials.gov/large-docs/87/NCT03888287/Prot_SAP_000.pdf